CLINICAL TRIAL: NCT00238108
Title: Melatonin Supplementation in Hypertensive Patients
Brief Title: Melatonin Supplements for Improving Sleep in Individuals With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT002713 (NIH); R21AT002713 (NIH)
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Sleep Disorders; Hypertension
Keywords: Sleep disorders; High blood pressure
MeSH Terms: conditions — Sleep Wake Disorders; Hypertension | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Melatonin (2,5 mg, by mouth, 1 per day, for 3-4 weeks)
  Interventions: Drug: Melatonin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 2,5 mg melatonin, by mouth, 1 per day, for 3-4 weeks
  Other Names: N-acetyl-5-methoxytryptamine
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of treatment with melatonin supplements in improving sleep in individuals with high blood pressure who are taking beta-blockers.

DETAILED DESCRIPTION:
Hypertension, or high blood pressure, is a condition in which an individual's blood pressure is higher than the normal level. It is estimated that one in three individuals in the United States has high blood pressure, though many do not know it because there are usually no symptoms. Uncontrolled hypertension may lead to stroke, heart attack, heart failure, or kidney failure. Beta-blockers are one class of drugs that have been developed to help lower blood pressure, and thereby decrease the risk for these serious problems. Beta-blockers also lower the levels of melatonin, a hormone that has a sleep-promoting effect. Many individuals who take beta-blockers for hypertension complain that they have trouble sleeping, which may be related to the beta-blockers' effect on melatonin levels. This study will evaluate the effectiveness of treatment with melatonin supplements in improving sleep in individuals with high blood pressure who are taking beta-blockers. In addition, the study will examine whether the melatonin supplements aid in lowering blood pressure.

Participants in this double-blind study will be randomly assigned to receive either melatonin supplements or placebo for the duration of the study. Participants will take part in two inpatient phases. Each inpatient stay will last 4 days and will be separated by 3 to 4 weeks. While in the clinic, participants' sleep patterns and core temperature will be recorded and plasma, saliva, and urine samples will be collected. Blood pressure will be measured before and after each inpatient stay, as well as at points during the stay. Throughout the study, participants' activity will be monitored by an accelerometer worn around the wrist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with uncomplicated hypertension
* Currently being treated with Atenolol (a beta-blocker)

Exclusion Criteria:

* History of medical illness other than essential hypertension
* Personal or family history of psychiatric illness
* Current use of any medication other than anti-hypertensive drugs
* Any recent travel across time zones
* History of working various shifts on an irregular basis

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank AJ Scheer, PhD, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Scheer FA, Van Montfrans GA, van Someren EJ, Mairuhu G, Buijs RM. Daily nighttime melatonin reduces blood pressure in male patients with essential hypertension. Hypertension. 2004 Feb;43(2):192-7. doi: 10.1161/01.HYP.0000113293.15186.3b. Epub 2004 Jan 19. PMID 14732734
- [Derived] Scheer FA, Morris CJ, Garcia JI, Smales C, Kelly EE, Marks J, Malhotra A, Shea SA. Repeated melatonin supplementation improves sleep in hypertensive patients treated with beta-blockers: a randomized controlled trial. Sleep. 2012 Oct 1;35(10):1395-402. doi: 10.5665/sleep.2122. PMID 23024438

RESULTS

PARTICIPANT FLOW:
Groups:
- Melatonin: Melatonin
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (6.9) | 56 (5.7) | 56 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality
Description: Sleep efficiency as measured by polysomnography (total time asleep as a percentage of the 8-hour sleep opportunity)
Time Frame: Measurement after 3 weeks of supplementation
Population: One subject was removed from analysis because of an unstable dose of prescription medication.
Measure: Mean (Standard Error); unit: % (% asleep during 8 hour opportunity)
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 7 | 8
% (% asleep during 8 hour opportunity) | 88.1 (2.7) | 80.5 (2.6)

2. Secondary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure as measured by 24-h ambulatory blood pressure monitoring
Time Frame: Measurement after 3 weeks of supplementation compared to baseline
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 7 | 8
mmHg | -0.2 (2.7) | -0.4 (2.7)

ADVERSE EVENTS:
Arm/Group | Melatonin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes